CLINICAL TRIAL: NCT04268355
Title: MINDFUL-PC for Portuguese Speakers Pilot #2 Study 2020 (Integrating Mindfulness Into the Patient-Centered Medical Home)
Brief Title: MINDFUL-PC for Portuguese Speakers Pilot Study 2020
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In order to ensure patients and research staff safety due to COVID-19 pandemic
Sponsor: Cambridge Health Alliance (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CambridgeHA; UH3AT009145 (NIH)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Depression; Anxiety Disorders; Stress Related Disorder; Adjustment Disorders; Chronic Illness
MeSH Terms: conditions — Depression; Anxiety Disorders; Adjustment Disorders; Chronic Disease | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: Single-arm, pre-post, non-randomized, unblinded pilot trial including up to 36 participants over 2 MTPC group cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindfulness Training for Primary Care (Experimental): Mindfulness Training for Primary Care (MTPC) is a primary care adaptation that includes core common Mindfulness-Based Intervention (MBI) elements integrated with novel mindfulness-oriented behavior change elements into a format that is adaptable to delivery in primary care health centers
  Interventions: Behavioral: Mindfulness Training for Primary Care

INTERVENTIONS:
Behavioral: Mindfulness Training for Primary Care — MTPC is a referral-based, insurance-reimbursable 8-week program delivered as group psychotherapy by Patient-Centered Medical Home-integrated behavioral clinicians or as an 8-week primary care group visit delivered by a primary care provider. MTPC groups are 2 hours for 8 weeks with a 7-hour weekend day of silent practice. MTPC emphasizes mindfulness-oriented skills for self-regulation, self-management of chronic illness, and health behavior change. All participants complete an action plan during Week 7. Participants are called every two weeks for the first eight weeks for 5-10 minute engagement calls which focus helping participants cultivate a relationship with study staff, giving participants a place to ask questions, and supporting participants in completing study visits.

SUMMARY:
The study evaluates the effects of the Mindfulness Training for Primary Care (MTPC) Portuguese-adapted version on heart rate variability during a demanding cognitive task. The study also evaluates the effects on mental health, quality of life, self-regulation and behavior outcomes. The study will also complete the MTPC cultural adaptation process for Brazilian culture.

DETAILED DESCRIPTION:
This single-arm, pre-post, non-randomized, unblinded, pilot trial evaluates the effects of Mindfulness Training for Primary Care (MTPC) Portuguese-adapted version on heart rate variability during a demanding cognitive task, i.e., Sustained Attention to Response Task (SART). Secondary aims are the following: 1) to measure pre/post outcomes for a) mental health (anxiety, depression, stress); b) quality of life; c) self-regulation (self-compassion, mindfulness, interoceptive awareness, difficulties in emotion regulation); and to determine the rate of d) chronic disease self-management action plan initiation; and 2) to complete the MTPC cultural adaptation for Brazilian culture through a) Satisfaction and Suggestions Survey; and b) Interviews of MTPC Group Leaders about their experience teaching the program Portuguese-adapted version.

ELIGIBILITY:
Inclusion Criteria:

* Current CHA patient with an enrolled CHA primary care doctor.
* CHA patients 18 years of age and older.
* Able to tolerate and participate in interviews and engage in all procedures.
* Diagnosis eligible to be covered by insurance for group visits (e.g., anxiety disorder, depression, stress disorders including adjustment disorder related to chronic illness, pain, insomnia, etc.).
* Must be able to fill out the study questionnaires on a computer or compatible mobile device.
* Must be willing to attend the two computer task sessions.
* Able to give written consent in Portuguese

Exclusion Criteria:

* Any cognitive impairment that precludes informed consent.
* Patients who, in the opinion of the Principal Investigator, pose an imminent risk of suicide or danger to self or others.
* Likelihood of potential incarceration such as a conviction or pending charges that may potentially result in imprisonment.
* Behaviors that may cause disruption to a mindfulness group.
* Patients with symptoms of psychosis, thought disorder, and/or severe mental illness, including schizophrenia, schizoaffective, bipolar disorder, or a current severe episode of major depressive disorder.
* Refusal of insurance to cover group psychotherapy treatment may lead to exclusion from participation in groups.
* Patients in their third trimester of pregnancy who foresee conflicts that preclude their commitment to completing all activities.
* Patients with highly unstable medical problems that put them at a high risk of hospitalization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
High-Frequency power (HF) - Heart Rate Variability (HRV) during Sustained Attention to Response Task (SART) last 5 minutes | Week 9
  High-Frequency power (HF) - Heart Rate Variability (HRV) during Sustained Attention to Response Task (SART) last 5 minutes will be measured using Biostamp nPoint® medical device. During SART participants complete a computerized test measuring sustained attention and response inhibition. They are asked to press a key in response to rapidly displayed integers (1-9) and withhold a response to a designated "no-go" integer.

SECONDARY OUTCOMES:
Root Mean Square of the Successive Differences (RMSSD) - Heart Rate Variability (HRV) during Sustained Attention to Response Task (SART) last 5 minutes | Week 9
  Root Mean Square of the Successive Differences (RMSSD) - Heart Rate Variability (HRV) during Sustained Attention to Response Task (SART) last 5 minutes will be measured using Biostamp nPoint® medical device. During SART participants complete a computerized test measuring sustained attention and response inhibition. They are asked to press a key in response to rapidly displayed integers (1-9) and withhold a response to a designated "no-go" integer.
Perceived Stress Scale (PSS-14) | Week 8
  The Perceived Stress Scale (PSS-14) (14 items) measures the degree to which situations in life are stressful. Items are designed to evaluate how overloaded, unpredictable, and uncontrollable one finds one's life. Each item is scored on a 5 point Likert scale from 0 (Never) to 4 (Very often).
Patient Reported Outcomes Measurement Information System - Anxiety Short Form (PROMIS-ASF) | Week 8
  The Patient Reported Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-ASF) is an 8-item scale used to assess patient-reported health status for anxiety. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Participants are asked to rate their experience of the item in the past seven days on a 5-point scale from 1 (Never) to 5 (Always).
Patient Reported Outcomes Measurement Information System - Depression Short Form (PROMIS-DSF) | Week 8
  The Patient Reported Outcomes Measurement Information System - Depression Short Form 8a (PROMIS-DSF) is an 8-item scale used to assess patient-reported health status for depression. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Participants are asked to rate their experience of the item in the past seven days on a 5-point scale from 1 (Never) to 5 (Always).

OTHER OUTCOMES:
High-Frequency power (HF) - Heart Rate Variability (HRV) during four 5-minute Sustained Attention to Response Task (SART) time blocks | Week 9
  High-Frequency power (HF) - Heart Rate Variability (HRV) during four 5-minute Sustained Attention to Response Task (SART) time blocks will be measured using Biostamp nPoint® medical device. During SART participants complete a computerized test measuring sustained attention and response inhibition. They are asked to press a key in response to rapidly displayed integers (1-9) and withhold a response to a designated "no-go" integer. Relationship between HF-HRV and SART performance will be evaluated and the effect of over time during the demanding SART task will also be evaluated.
Root Mean Square of the Successive Differences (RMSSD) - Heart Rate Variability (HRV) during four 5-minute Sustained Attention to Response Task (SART) time blocks | Week 9
  Root Mean Square of the Successive Differences (RMSSD) - Heart Rate Variability (HRV) during four 5-minute Sustained Attention to Response Task (SART) time blocks will be measured using Biostamp nPoint® medical device. During SART participants complete a computerized test measuring sustained attention and response inhibition. They are asked to press a key in response to rapidly displayed integers (1-9) and withhold a response to a designated "no-go" integer. Relationship between RMSSD and SART performance will be evaluated and the effect of over time during the demanding SART task will also be evaluated.
Action Plan Initiation Survey (APIS-5) | Week 9
  Patient self-reported Action Plan Initiation is based on two-item in the APIS-5 self-report survey in which patients are asked to list their action plan SMART goal, if they met the goal and how much control they had over meeting the goal. The main outcome is a single-item response determining whether they met or did not meet the goal using a 7-point Likert scale (ranging from 1-7) with scores >=5 representing self-reported initiation of the goal.
World Health Organization Quality of Life- BREF (WHOQOL-BREF) | Week 8
  The World Health Organization has developed a quality of life instrument, the WHOQOL, which captures many subjective aspects of quality of life. The WHOQOL-BREF is a WHOQOL shorter version, comprises 26 items that produces scores for four domains related to quality of life: physical health, psychological, social relationships and environment. It also includes one facet on overall quality of life and general health.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Week 8
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item self-report scale designed to assess multiple aspects of interoception and interoceptive awareness. The 6 point Likert scale (ranging from 0-6) assesses 8 aspects of interoceptive awareness: noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. Subscales are averaged, and a higher total score represents a better outcome.
Difficulty in Emotion Regulation Scale (DERS) | Week 8
  The Difficulties in Emotion Regulation (DERS) Scale is a 36-item self-report scale designed to assess emotional dysregulation using a 5 point Likert scale. The scale assesses 6 aspects of emotional dysregulation: non-acceptance of emotional responses, difficulties engaging in goal directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Subscales are summed and a lower total score represents a better outcome.
Five Facet Mindfulness Questionnaire (FFMQ) | Week 8
  The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item scale that examines five factors that represent aspects of the current empirical conception of mindfulness. These five facets include: "observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience." Participants rate their degree of agreement with each of the items on a Likert-type scale ranging from 1 (Never or very rarely true) to 5 (Very often or always true), with higher scores indicating higher experience of mindfulness.
Self-Compassion Scale (SCS) | Week 8
  The Self-Compassion Scale is composed by 26 items measuring six components of self-compassion: self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification.The items are rated on a five-point response scale ranging from 1 (almost never) to 5 (almost always).
Satisfaction Survey | Week 8
  Satisfaction Survey is an 18-item survey contains two parts. First is a series of 12 questions scored on a 5-point Likert scale from 1 (Strongly Disagree/Poor) to 5 (Strongly Agree/Excellent), with statements such as "I found this program helpful." Next is a series of six open-ended questions in which patients enter a written response to statements including "The most important thing I learned during this program."
Suggestions Survey | Week 8
  The Suggestions Survey consist of 4 questions focusing on the intervention cultural aspects.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gawande R, To MN, Pine E, Griswold T, Creedon TB, Brunel A, Lozada A, Loucks EB, Schuman-Olivier Z. Mindfulness Training Enhances Self-Regulation and Facilitates Health Behavior Change for Primary Care Patients: a Randomized Controlled Trial. J Gen Intern Med. 2019 Feb;34(2):293-302. doi: 10.1007/s11606-018-4739-5. Epub 2018 Dec 3. PMID 30511291
- [Background] Gawande R, Pine E, Griswold T, Creedon T, Vallejo Z, Rosenbaum E, Lozada A, Schuman-Olivier Z. Insurance-Reimbursable Mindfulness for Safety-Net Primary Care Patients: A Pilot Randomized Controlled Trial. Mindfulness (N Y). 2019 Sep;10(9):1744-1759. doi: 10.1007/s12671-019-01116-8. Epub 2019 Mar 18. PMID 32042349
- [Derived] Trombka M, Creedon TB, Demarzo M, Cuoco LT, Smith L, Oxnard AC, Rozembaque AT, Hirayama MS, Moreno NB, Comeau A, Gawande R, Griswold T, Cook BL, Rocha NS, Schuman-Olivier Z. Mindfulness Training for Primary Care for Portuguese-Speaking Immigrants: A Pilot Study. Front Psychiatry. 2021 Sep 9;12:664381. doi: 10.3389/fpsyt.2021.664381. eCollection 2021. PMID 34566708